CLINICAL TRIAL: NCT04120363
Title: A Randomized, Double-blind, Placebo Controlled Trial of Testosterone Undecanoate for Optimizing Physical and Cognitive Performance During Military Operations (OPS II)
Brief Title: Trial of Testosterone Undecanoate for Optimizing Performance During Military Operations
Acronym: OPS II
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency); United States Department of Defense (U.S. Federal Agency); University of Arkansas (Other)
Responsible Party: Principal Investigator, Jennifer C. Rood, Principal Investigator, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PBRC 2019-017; W81XWH19C0162 (Other Grant/Funding Number: USA MED RESEARCH ACQ ACTIVITY); W81XWH19D0010 (Other Grant/Funding Number: USA MED RESEARCH ACQ ACTIVITY)
Record Dates: First submitted 2019-10-04; First posted 2019-10-09 (Actual); Results first posted 2022-10-07 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-09

CONDITIONS: Caloric Restriction; Exercise; Sleep
Keywords: testosterone; anabolism; muscle mass; military operational stress
MeSH Terms: conditions — Motor Activity | interventions — testosterone undecanoate; Testosterone Propionate; Sesame Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): single intramuscular injection of 750 mg sesame oil solution on Day 8
  Interventions: Drug: Sesame Oil
- Testosterone (Experimental): single intramuscular injection of 750 mg testosterone undecanoate on Day 8
  Interventions: Drug: Testosterone Undecanoate

INTERVENTIONS:
Drug: Testosterone Undecanoate — single intramuscular injection of 750 mg testosterone undecanoate
  Other Names: Aveed
  Arms: Testosterone
Drug: Sesame Oil — single intramuscular injection of 750 mg sesame oil solution
  Arms: Placebo

SUMMARY:
The objective of this study is to determine the effects of a single dose of testosterone undecanoate during and in recovery from simulated operational stress.

DETAILED DESCRIPTION:
This is a double-blind, randomized, placebo controlled trial in 32 physically active men exposed to 20 complete days (days 8-27) of simulated operational stress followed by 20 complete days of recovery (days 29-48). After completing baseline testing (Phase 1), participants will be randomized to receive either a single intramuscular injection of testosterone undecanoate or an isovolumetric placebo (Day 8). The 20-day simulated operational stress (Phase 2) will be highly controlled (live-in study) and consist of 4 successive cycles of undulating stress, starting with 2 consecutive days of low stress followed by 3 consecutive days of high stress. Low- and high-stress days will result from low and high militarily-relevant exercise-induced energy expenditures, adequate and restricted sleep (8 hours vs. 4 hours daily), and diet restriction to produce energy deficits. After completing Phase 2, participants will be released to resume their habitual physical activity routines and will be provided a controlled diet to consume (Phase 3), to assess recovery from sustained, severe operational stress.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 18-35 years
* Ability to understand verbal or written instructions/testing materials in English
* Physically active (as determined by accelerometry and review of a physical activity log)
* Not taking any prescription medications and/or willing to refrain from all medication use prior to and throughout the entire study period, unless provided/approved by the study physician
* Willing to refrain from alcohol, smoking, e-cigarettes or use of any nicotine product, caffeine, and dietary supplement use throughout the entire study period
* Willing to live on the Pennington Biomedical Research Center inpatient unit for 20 consecutive days
* Meets age-specific US Army body composition standards according to Army Regulation 600-9, which includes estimates of percent body fat based on height, weight, and circumference measures (neck and waist)
* Total testosterone concentration is within the normal physiological range (300-1,000 ng/dL)

Exclusion Criteria:

* Musculoskeletal injuries that compromise exercise capability
* Diagnosed cardiometabolic disorders (i.e., hypertension, hyperlipidemia, kidney disease, diabetes, etc.)
* Allergies or intolerance to foods, vegetarian practices, or history of complications with lidocaine
* Anabolic steroid, human growth hormone, or nutritional testosterone precursor-like supplement use within the past 6 months
* Will not refrain from smoking (any nicotine product), alcohol, caffeine, or any other dietary supplement during the study
* Adults unable to consent
* Women
* Prisoners
* Sedentary or engages in insufficient quantities of physical activity per week (aerobic and/or resistance training as determined by accelerometry and review of a physical activity log)
* Exceeds age-specific US Army body composition standards according to Army Regulation 600-9
* Previous history of kidney stones unless otherwise approved by the medical investigator
* Systolic blood pressure > 150 or diastolic blood pressure > 95 mmHg
* Previous history of breast or prostate cancer
* Previous history of Chronic Obstructive Pulmonary Disease or Obstructive Sleep Apnea
* Prostate-Specific Antigen (PSA) > 3ng/ml, Hematocrit > 50%, or positive urine drug screening
* Based on the investigative team's clinical judgment, a subject may not be appropriate for participation in the study

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2021-07-08 (Actual); Study Completion 2021-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer C Rood, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lowe AC, Niclou A, Varanoske AN, Harris MN, Hebert C, Johannsen NM, Heymsfield SB, Greenway FL, Margolis LM, Lieberman HR, Beyl RA, Ferrando AA, Pasiakos SM, Rood JC. Exercise Heart Rate Variability Suggests Parasympathetic Hyperactivity during Simulated Military Operations Irrespective of Testosterone Administration. Med Sci Sports Exerc. 2025 Sep 1;57(9):1979-1987. doi: 10.1249/MSS.0000000000003743. Epub 2025 Apr 25. PMID 40279652
- [Derived] Varanoske AN, Harris MN, Hebert C, Johannsen NM, Heymsfield SB, Greenway FL, Ferrando AA, Rood JC, Pasiakos SM. Bioelectrical impedance phase angle is associated with physical performance before but not after simulated multi-stressor military operations. Physiol Rep. 2023 Mar;11(6):e15649. doi: 10.14814/phy2.15649. PMID 36949577
- [Derived] Wong MC, Bennett JP, Leong LT, Tian IY, Liu YE, Kelly NN, McCarthy C, Wong JMW, Ebbeling CB, Ludwig DS, Irving BA, Scott MC, Stampley J, Davis B, Johannsen N, Matthews R, Vincellette C, Garber AK, Maskarinec G, Weiss E, Rood J, Varanoske AN, Pasiakos SM, Heymsfield SB, Shepherd JA. Monitoring body composition change for intervention studies with advancing 3D optical imaging technology in comparison to dual-energy X-ray absorptiometry. Am J Clin Nutr. 2023 Apr;117(4):802-813. doi: 10.1016/j.ajcnut.2023.02.006. Epub 2023 Feb 14. PMID 36796647
- [Derived] Varanoske AN, Harris MN, Hebert C, Howard EE, Johannsen NM, Heymsfield SB, Greenway FL, Margolis LM, Lieberman HR, Church DD, Ferrando AA, Rood JC, Pasiakos SM. Effects of testosterone undecanoate on performance during multi-stressor military operations: A trial protocol for the Optimizing Performance for Soldiers II study. Contemp Clin Trials Commun. 2021 Jul 3;23:100819. doi: 10.1016/j.conctc.2021.100819. eCollection 2021 Sep. PMID 34278044

RESULTS

PARTICIPANT FLOW:
Period: Phase 1
Arm/Group | Testosterone | Placebo
Started | 16 | 18
Completed | 16 | 18
Not Completed | 0 | 0
Period: Phase 2
Arm/Group | Testosterone | Placebo
Started | 16 | 18
Completed | 16 | 16
Not Completed | 0 | 2
Period: Phase 3
Arm/Group | Testosterone | Placebo
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Testosterone | Placebo | Total
Number analyzed (Participants) | 16 | 18 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.9 (4.4) | 26.2 (4.5) | 26.5 (4.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 16 | 18 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 13 | 16 | 29
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 5 | 8
  White | 11 | 12 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Body Mass [Mean (Standard Deviation); unit: kg] | 76.5 (14.7) | 77.5 (10.2) | 77.1 (12.3)
Height [Mean (Standard Deviation); unit: cm] | 177.1 (8.1) | 176.3 (5.3) | 176.7 (6.7)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 24.3 (3.8) | 24.9 (2.7) | 24.6 (3.2)

OUTCOME MEASURES:

1. Primary Outcome: Load Carriage Time
Description: A load carriage time trial (a militarily relevant aerobic performance assessment) was conducted near the end of each study phase to assess aerobic performance.
Time Frame: Day 5 (Phase 1), Day 26 (Phase 2), Day 47 (Phase 3)
Population: 2 participants in the placebo group dropped out of the study during Phase 2
Measure: Least Squares Mean (Standard Error); unit: min
Arm/Group | Testosterone | Placebo
Number analyzed (Participants) | 16 | 18
min
  2.5 mile time, Phase 1 | 45.21 (2.01) | 41.58 (1.94)
  2.5 mile time, Phase 2: number analyzed (Participants) | 16 | 16
  2.5 mile time, Phase 2 | 50.95 (2.01) | 47.15 (1.99)
  2.5 mile time, Phase 3: number analyzed (Participants) | 16 | 16
  2.5 mile time, Phase 3 | 44.31 (2.07) | 39.34 (2.12)

2. Secondary Outcome: Body Composition
Description: A four-compartment (4C) model factoring in body mass, body volume, total body water, and bone mineral content was used to calculate fat-free body mass and fat mass at the end of each study phase.
Time Frame: Day 7 (Phase 1), Day 28 (Phase 2), Day 49 (Phase 3)
Population: 2 participants in the placebo group dropped out of the study during Phase 2
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Testosterone | Placebo
Number analyzed (Participants) | 16 | 18
kg
  Fat-free Mass at end of Phase 1 | 59.2 (2.0) | 59.8 (2.1)
  Fat-free Mass at end of Phase 2: number analyzed (Participants) | 16 | 16
  Fat-free Mass at end of Phase 2 | 59.6 (2.0) | 57.9 (2.1)
  Fat-free Mass at end of Phase 3: number analyzed (Participants) | 16 | 16
  Fat-free Mass at end of Phase 3 | 59.5 (2.0) | 59.6 (2.1)
  Fat Mass at end of Phase 1 | 17.3 (1.5) | 17.5 (1.6)
  Fat Mass at end of Phase 2: number analyzed (Participants) | 16 | 16
  Fat Mass at end of Phase 2 | 13.0 (1.5) | 14.4 (1.6)
  Fat Mass at end of Phase 3: number analyzed (Participants) | 16 | 16
  Fat Mass at end of Phase 3 | 15.1 (1.5) | 15.5 (1.6)

3. Primary Outcome: Vertical Jump Height
Description: Lower-body peak power was assessed near the end of each phase using a vertical jump test.
Time Frame: Day 4 (Phase 1), Day 25 (Phase 2), Day 46 (Phase 3)
Population: 2 participants in the placebo group dropped out of the study during Phase 2
Measure: Least Squares Mean (Standard Error); unit: cm
Arm/Group | Testosterone | Placebo
Number analyzed (Participants) | 16 | 18
cm
  Vertical Jump Height, Phase 1 | 54.5 (2.5) | 53.6 (2.4)
  Vertical Jump Height, Phase 2: number analyzed (Participants) | 16 | 16
  Vertical Jump Height, Phase 2 | 49.1 (2.5) | 50.0 (2.5)
  Vertical Jump Height, Phase 3: number analyzed (Participants) | 16 | 16
  Vertical Jump Height, Phase 3 | 54.0 (2.5) | 50.5 (2.5)

4. Primary Outcome: Total Mass Lifted
Description: A 3-repetition maximum deadlift assessed muscular strength, endurance, and explosive power near the end of each study phase.
Time Frame: Day 4 (Phase 1), Day 25 (Phase 2), Day 46 (Phase 3)
Population: 2 participants in the placebo group dropped out of the study during Phase 2
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Testosterone | Placebo
Number analyzed (Participants) | 16 | 18
kg
  Total Mass Lifted, Phase 1 | 127.4 (7.4) | 127.9 (7.0)
  Total Mass Lifted, Phase 2: number analyzed (Participants) | 16 | 16
  Total Mass Lifted, Phase 2 | 122.7 (7.4) | 119.0 (7.2)
  Total Mass Lifted, Phase 3: number analyzed (Participants) | 16 | 16
  Total Mass Lifted, Phase 3 | 126.7 (7.7) | 129.8 (7.2)

5. Primary Outcome: Wingate Peak Power
Description: Anaerobic capacity was assessed using a Wingate anaerobic cycle test near the end of each study phase.
Time Frame: Day 4 (Phase 1), Day 25 (Phase 2), Day 46 (Phase 3)
Population: 2 participants in the placebo group dropped out of the study during Phase 2
Measure: Least Squares Mean (Standard Error); unit: W
Arm/Group | Testosterone | Placebo
Number analyzed (Participants) | 16 | 18
W
  Wingate peak power, absolute, Phase 1 | 879.4 (49.6) | 837.8 (49.6)
  Wingate peak power, absolute, Phase 2: number analyzed (Participants) | 16 | 16
  Wingate peak power, absolute, Phase 2 | 753.8 (49.6) | 736.0 (49.6)
  Wingate peak power, absolute, Phase 3: number analyzed (Participants) | 16 | 16
  Wingate peak power, absolute, Phase 3 | 821.8 (49.6) | 790.8 (49.6)

6. Primary Outcome: Peak Aerobic Capacity
Description: Peak aerobic capacity was measured via treadmill VO2peak near the end of each study phase.
Time Frame: Day 4 (Phase 1), Day 25 (Phase 2), Day 46 (Phase 3)
Population: 2 participants in the placebo group dropped out of the study during Phase 2
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | Testosterone | Placebo
Number analyzed (Participants) | 16 | 18
L/min
  VO2peak, absolute, Phase 1 | 3.22 (0.15) | 3.28 (0.14)
  VO2peak, absolute, Phase 2: number analyzed (Participants) | 16 | 16
  VO2peak, absolute, Phase 2 | 3.13 (0.15) | 3.20 (0.14)
  VO2peak, absolute, Phase 3: number analyzed (Participants) | 16 | 16
  VO2peak, absolute, Phase 3 | 3.29 (0.15) | 3.44 (0.14)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the time of the screening visit until study completion, up to 4 months.
Arm/Group | Testosterone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/18
Other Adverse Events (participants affected / at risk) | 15/16 | 16/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Testosterone (N=16) | Placebo (N=18)
Cardiovascular issues (Vascular disorders) | 1 (1) | 1 (1)
Dermatologic issues (Skin and subcutaneous tissue disorders) | 13 (25) | 14 (26)
Gastrointestinal issues (Gastrointestinal disorders) | 7 (9) | 3 (5)
Genitourinary issues (Renal and urinary disorders) | 1 (1) | 0 (0)
Musculoskeletal issues (Musculoskeletal and connective tissue disorders) | 15 (54) | 16 (40)
Neurological issues (Nervous system disorders) | 5 (7) | 4 (6)
Nonspecific issues (General disorders) | 6 (8) | 5 (5)
Oral complaints (General disorders) | 4 (4) | 2 (2)
Respiratory issues (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 4 (4)
Special senses issues (General disorders) | 3 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-08-24): https://cdn.clinicaltrials.gov/large-docs/63/NCT04120363/Prot_SAP_000.pdf
  • Informed Consent Form (2020-08-24): https://cdn.clinicaltrials.gov/large-docs/63/NCT04120363/ICF_001.pdf